CLINICAL TRIAL: NCT01553604
Title: Influence of Dressing Wear Time on Skin Colonization After Breast Augmentation With Prosthesis: a Randomized Controlled Trial
Brief Title: Dressing Wear Time After Breast Augmentation With Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Francescato Veiga (Other)
Responsible Party: Sponsor-Investigator, Daniela Francescato Veiga, Professor, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Micro02
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Surgical Site Infection
Keywords: breast prosthesis implantation; bandages; skin colonization; surgical site infection; augmentation mammaplasty; dressing wear time
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postoperative day 6 (Experimental): Dressing is removed on the sixth postoperative day
  Interventions: Procedure: augmentation mammaplasty
- Postoperative day 1 (Experimental): Dressing is removed on the first postoperative day
  Interventions: Procedure: augmentation mammaplasty

INTERVENTIONS:
Procedure: augmentation mammaplasty — Dressing is removed on the first postoperative day
  Arms: Postoperative day 1
Procedure: augmentation mammaplasty — Dressing is removed on the 6th postoperative day
  Arms: Postoperative day 6

SUMMARY:
This study was designed to determine whether the duration of dressing wear following augmentation mammaplasty influence skin colonization and eventually surgical site infections rates.

DETAILED DESCRIPTION:
Augmentation mammaplasty is currently one of the most performed plastic surgery procedures. It is a clean operation, and surgical site infection (SSI) rates are low. However, a SSI, since a minor one, leads to the failure of the procedure. Thus, minimizing SSI risks is imperative.

The Centers for Disease Control and Prevention (CDC) provides recommendations concerning prevention of SSI.No recommendation is offered for some practices, either because there is a lack of consensus regarding their efficacy or because of the available scientific evidence is insufficient to support their adoption.

CDC´s "Guideline for Prevention of Surgical Site Infection" recommends protecting with a sterile dressing for 24 to 48 hours an incision that has been closed primarily. There is no recommendation to cover the incision beyond 48 hours. One major risk factor for SSI is the presence of bacteria at surgical site.Thus, this trial was designed to verify the influence of dressing wear time on skin colonization.

ELIGIBILITY:
Inclusion Criteria:

* candidate to breast prosthesis implantation
* body mass index under 30Kg/m2

Exclusion Criteria:

* pregnancy, delivery or breast feeding during the last 12 months
* body mass index over 30Kg/m2
* breast cancer history
* previous breast surgery
* hard smoking

Ages: 18 Months to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
skin colonization | 6 days postoperatively
  skin colonization will be measured through semi-quantitative cultures of samples collected pre-dressing and on 6th postoperative day.

SECONDARY OUTCOMES:
surgical site infection | 30 days postoperatively
  Surgical site infection will be assessed weekly, for 30 days. CDC´s criteria and definitions will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela F Veiga, MD, PhD, Study Director — Universidade Federal de São Paulo; Joel Veiga-Filho, MD, PhD, Principal Investigator — Universidade do Vale do Sapucaí; Lydia M Ferreira, MD, PhD, Study Chair — Universidade Federal de São Paulo; Denise A Mendes, MD, PhD, Principal Investigator — Universidade Federal de São Paulo
Locations (1):
- Hospital das Clínicas Samuel Libanio, Pouso Alegre, Minas Gerais, Brazil

REFERENCES:
- [Background] Mendes Dde A, Veiga DF, Veiga-Filho J, Fonseca FE, de Paiva LF, Novo NF, Loyola AB, Ferreira LM. Application time for postoperative wound dressing following breast augmentation with implants: study protocol for a randomized controlled trial. Trials. 2015 Jan 27;16:19. doi: 10.1186/s13063-014-0529-5. PMID 25623237
- [Result] Mendes DA, Veiga DF, Veiga-Filho J, Loyola ABAT, Paiva LF, Novo NF, Sabino-Neto M, Ferreira LM. Influence of dressing application time after breast augmentation on cutaneous colonization: A randomized clinical trial. J Plast Reconstr Aesthet Surg. 2018 Jun;71(6):906-912. doi: 10.1016/j.bjps.2018.01.021. Epub 2018 Feb 21. PMID 29475792